CLINICAL TRIAL: NCT00460317
Title: A Phase 3, Multicenter, Randomized, Placebo-Controlled, Double-Blind Trial of AMG 706 in Combination With Paclitaxel and Carboplatin for Advanced Non-small Cell Lung Cancer.
Brief Title: MONET1-MOtesanib NSCLC Efficacy and Tolerability Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Amgen discontinued the development of AMG706 because 20050201 did not meet its primary objective.
Sponsor: Amgen (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20050201
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: lung; cancer; chemotherapy; paclitaxel; carboplatin; placebo; angiogenesis; VEGF; multi kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — motesanib diphosphate; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B (Placebo Comparator): All subjects on this treatment arm will receive a standard paclitaxel and carboplatin chemotherapy regimen (paclitaxel 200mg/m2 and carboplatin at AUC of 6mg/mL x min by Calvert formula) on day 1 of each 3 week cycle + - 3 days for a maximum of 6 cycles and placebo 125mg QD orally
  Interventions: Drug: placebo; Drug: paclitaxel; Drug: carboplatin
- Arm A (Active Comparator): All subjects on this treatment arm will receive a standard paclitaxel and carboplatin chemotherapy regimen (paclitaxel 200mg/m2 and carboplatin at AUC of 6mg/mL x min by Calvert formula) on day 1 of each 3 week cycle + - 3 days for a maximum of 6 cycles and AMG 706 125mg QD orally.
  Interventions: Drug: AMG 706; Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: AMG 706 — 125 mg QD orally every day
  Arms: Arm A
Drug: placebo — 125 mg QD orally every day
  Arms: Arm B
Drug: paclitaxel — 200mg/m2 on day 1 of each 3 week cycle +/- 3 days for a max of 6 cycles
Drug: carboplatin — AUC of 600mg/mL x min by Calvert formula on day 1 of each 3 week cycle +/- 3 days for a max of 6 cycles

SUMMARY:
To determine if treatment with AMG 706 (motesanib diphosphate) in combination with paclitaxel and carboplatin improves overall survival compared to treatment with placebo in combination with paclitaxel and carboplatin in subjects with advanced non-squamous NSCLC and in subjects with adenocarcinoma histology (adenocarcinoma subpopulation).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable stage 111B with pericardial or pleural effusion or stage IV or recurrent non squamous NSCLC.
* Measurable or non-measurable disease per modified RECIST criteria
* ECOG performance status of 0 or 1
* Life expectancy of greater than or equal to 3 months as documented by the investigator
* ability to take oral medications
* competency to give written informed consent
* able to start protocol directed therapy within 7 days from date of randomization
* Hematological function, as follows:
* Absolute neutrophil count (ANC) > = 1.5 x 109/L
* Platelet count > = 100 x 109/L and < = 850 x 109/L
* Hemoglobin > =9 g/dL
* Renal function, as follows:
* Creatinine clearance > 40 mL/min (calculated by Cockcroft Gault formula)
* Urinary protein quantitative value of < = 30 mg in urinalysis or < = 1+ on dipstick unless quantitative protein is < 500 mg in a 24 hour urine sample
* Hepatic function, as follows:
* Aspartate aminotransferase (AST) < =2.5 x upper limit of normal (ULN) OR AST < 5 x ULN if liver metastases are present
* Alanine aminotransferase (ALT) < =2.5 x ULN OR ALT < 5 x ULN if liver metastases are present
* Alkaline phosphatase < = 2.0 x ULN OR alkaline phosphatase < 5 x ULN if liver or bone metastases are present
* Total bilirubin < 1.5 x ULN OR total bilirubin < 3 X ULN if subject has UGT1A1 promoter polymorphism (ie, Gilbert syndrome) confirmed by genotyping or Invader UGT1A1 Molecular Assay prior to randomization Partial thromboplastin (PTT) or activated partial thromboplastin time (aPTT) < = 1 x ULN and international normalized ratio (INR) < = 1.5 x ULN

Exclusion Criteria:

* Subjects with adenosquamous histology or an unclear histology subtype (eg, not otherwise specified) containing greater than 10% squamous cells
* untreated or symptomatic central nervous system metastases. Subjects with a history of brain metastases are eligible if definitive therapy has been administered (surgery and/or radiation therapy), there is no planned treatment for brain metastases, and the subject is clinically stable and is off corticosteroids for at least 2 weeks prior to randomization.
* Prior chemotherapy as follows: Any prior chemotherapy for advanced non squamous NSCLC
* Any prior adjuvant chemotherapy for non squamous NSCLC within 52 weeks prior to randomization. Adjuvant chemotherapy completed > 52 weeks prior to randomization is permitted. Any prior chemoradiation for locally advanced stage III disease.
* Prior (within 30 days of randomization) yellow fever vaccination.
* Central (chest) radiation therapy within 28 days prior to randomization, radiation therapy within 14 days prior to randomization for peripheral lesions.
* History of pulmonary hemorrhage or gross hemoptysis (approximately 3 mL of bright red blood or more) within 6 months prior to randomization.
* Prior targeted therapies, including but not limited to:
* AMG 706, inhibitors of VEGF (eg, SU5416, SU6668, ZD6474, SU11248, PTK787, AZD2171, AEE 788, sorafenib, bevacizumab), or EGFr (eg, panitumumab, cetuximab, gefitinib, erlotinib).
* Known history of allergy or hypersensitivity reaction to paclitaxel or carboplatin.
* Any anticoagulation therapy within 7 days prior to randomization. The use of low-dose warfarin [ < = 2 mg daily] or low molecular weight heparin or heparin flushes for prophylaxis against central venous catheter thrombosis is allowed.
* History of arterial or venous thrombosis within 12 months prior to randomization.
* History of bleeding diathesis or bleeding within 14 days prior to randomization.
* Peripheral neuropathy > grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
* Clinically significant cardiac disease within 12 months of randomization, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, percutaneous transluminal coronary angioplasty/stent, congestive heart failure, or ongoing arrhythmias requiring medication.
* History of other primary cancer unless: Curatively resected non melanomatous skin cancer. Curatively treated cervical carcinoma in situ. Other primary solid tumor curatively treated with no known active disease present and no curative treatment administered for the last 3 years
* Any kind of disorder that compromises the ability of the subject to comply with the study procedures.
* Open wound, ulcer or fracture.
* Uncontrolled hypertension as defined by resting blood pressure > 150/90 mm Hg. Antihypertensive medications are allowed if the subject is stable on their current dose at the time of randomization.
* Surgery:
* Major surgical procedures within 28 days prior to randomization
* Minor surgical procedures within 14 days prior to randomization
* Failure to recover from prior surgery
* Placement of a central venous access device (including ports and tunneled or non-tunneled catheters) within 7 days prior to randomization
* Planned elective surgery while on study treatment
* Core needle biopsy within 7 days prior to randomization
* Not recovered from all previous therapies (ie, radiation, surgery and medications). Adverse events related to previous therapies must be CTCAE grade < = 1 at screening or returned to the subject's baseline prior to their most recent previous therapy.
* Participation in therapeutic clinical trials or currently receiving other investigational treatment(s) within 30 days prior to randomization.
* Pregnant (eg, positive HCG test-serum or urine) or breast feeding woman.
* Any subject not consenting to use adequate contraceptive precautions (eg, hormonal, barrier or abstinence) during the course of the study and for 6 months after the last treatment.
* Known to be human immunodeficiency virus (HIV), hepatitis B surface antigen or hepatitis C positive.
* Known chronic hepatitis.
* Active infection requiring systemic treatment or any uncontrolled infection < = 14 days prior to randomization.
* History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results.
* Previously randomized to this study.
* Not available for follow-up assessments or unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1450 (Actual)
Dates: Start 2007-07; Primary Completion 2011-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Overall survival time. Time from randomization to death. Subjects who have not died while on study or are lost to follow up will be censored at their last contact date. | Not able to be measured

SECONDARY OUTCOMES:
Duration of response (calculated for only those subjects who respond) | Time from first objective tumour response to objective disease progression or death due to any cause.
Pharmacokinetics of AMG 706 when administered in combination with paclitaxel and carboplatin. | Throughout the duration the patient is in the study.
Association of AMG 706 treatment-induced PlGF increase with OS in subjects with non-squamous NSCLC and in subjects with adenocarcinoma histology | Overall survival time in the PlGF analysis set
Evaluation of OS, PFS, AMG 706 treatment-induced PlGF increase association with OS, ORR (only in subjects with measurable disease) and duration of response in subjects with non-squamous, non-adenocarcinoma histology | OS, ORR and duration of response in the PlGF analysis set
Evaluation of the pharmacokinetics of AMG 706 and metabolites when administered with paclitaxel and carboplatin (in approximately 250 subjects at selected centers) | Carboplatin PK samples drawn from subjects at Cycle 3 and Cycle 5
Safety and tolerability of AMG 706 in combination with paclitaxel and carboplatin compared to placebo in combination with paclitaxel and carboplatin in subjects with non-squamous NSCLC histology and in subjects with adenocarcinoma histology. | Throughout the duration the patient is in the study
Progression free survival time: Subjects who have not progressed or died on study will be censored at their last evaluable assessment date. | Time from randomization to objective disease progression or death due to any cause
Objective tumour response rate (complete and partial response) according to modified RECIST criteria in subjects with measurable disease at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Scagliotti GV, Vynnychenko I, Park K, Ichinose Y, Kubota K, Blackhall F, Pirker R, Galiulin R, Ciuleanu TE, Sydorenko O, Dediu M, Papai-Szekely Z, Banaclocha NM, McCoy S, Yao B, Hei YJ, Galimi F, Spigel DR. International, randomized, placebo-controlled, double-blind phase III study of motesanib plus carboplatin/paclitaxel in patients with advanced nonsquamous non-small-cell lung cancer: MONET1. J Clin Oncol. 2012 Aug 10;30(23):2829-36. doi: 10.1200/JCO.2011.41.4987. Epub 2012 Jul 2. PMID 22753922
- [Background] Bass MB, Yao B, Hei YJ, Ye Y, Davis GJ, Davis MT, Kaesdorf BA, Chan SS, Patterson SD. Challenges in developing a validated biomarker for angiogenesis inhibitors: the motesanib experience. PLoS One. 2014 Oct 14;9(10):e108048. doi: 10.1371/journal.pone.0108048. eCollection 2014. PMID 25314641
- [Background] Novello S, Scagliotti GV, Sydorenko O, Vynnychenko I, Volovat C, Schneider CP, Blackhall F, McCoy S, Hei YJ, Spigel DR. Motesanib plus carboplatin/paclitaxel in patients with advanced squamous non-small-cell lung cancer: results from the randomized controlled MONET1 study. J Thorac Oncol. 2014 Aug;9(8):1154-61. doi: 10.1097/JTO.0000000000000227. PMID 25157768
- [Derived] Kubota K, Ichinose Y, Scagliotti G, Spigel D, Kim JH, Shinkai T, Takeda K, Kim SW, Hsia TC, Li RK, Tiangco BJ, Yau S, Lim WT, Yao B, Hei YJ, Park K. Phase III study (MONET1) of motesanib plus carboplatin/paclitaxel in patients with advanced nonsquamous nonsmall-cell lung cancer (NSCLC): Asian subgroup analysis. Ann Oncol. 2014 Feb;25(2):529-36. doi: 10.1093/annonc/mdt552. Epub 2014 Jan 13. PMID 24419239
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com